CLINICAL TRIAL: NCT03018106
Title: Ospemifene Versus Conjugated Estrogens in the Treatment of Postmenopausal Sexual Dysfunction
Brief Title: Ospemifene vs. Conjugated Estrogens in the Treatment of Postmenopausal Sexual Dysfunction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Obstacles with recruitment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Gina Northington, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00088077
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-11

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Female sexual disorder; Aging; Menopause; Obstetrics/Gynecology; Female urogenital disorder
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Ospemifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ospemifene (Experimental): Women randomized to this arm will receive 60mg oral ospemifene, taken daily, for 12 weeks
  Interventions: Drug: Ospemifene
- Estrogen (Active Comparator): Women randomized to this arm will receive 0.5mg vaginal conjugated estrogens, placed vaginally twice per week, for 12 weeks
  Interventions: Drug: Vaginal conjugated estrogens

INTERVENTIONS:
Drug: Ospemifene — Ospemifene is a selective estrogen receptor modulator (SERM), and it is the only SERM approved in the United States to treat moderate to severe dyspareunia associated with VVA. It is an oral medication that is taken as a 60mg tablet once daily. Food intake increases its absorption by 2 to 3-fold, and this is not impacted by the fat or calorie content of the food. It is metabolized primarily in the liver, and is excreted in feces.
  Other Names: Osphena
  Arms: Ospemifene
Drug: Vaginal conjugated estrogens — Conjugated estrogens are a mixture of several different estrogen salts derived from natural sources and blended to approximate the composition of estrogens in the urine of pregnant horses. The main components are sodium estrone sulphate and sodium equilin sulfate. Vaginal estrogen is considered the medication of choice for treating vulvovaginal atrophy (VVA).
  Other Names: Premarin Vaginal Cream
  Arms: Estrogen

SUMMARY:
Vulvovaginal atrophy (VVA) is a condition that impacts up to 60% of the growing postmenopausal female population, and the most common symptom is dyspareunia. Vaginal estrogen is the most common treatment for VVA, but it only marginally improves overall sexual function, and many women and clinicians avoid using it because of the risks of exogenous estrogen use during menopause. Ospemifene is a non-estrogen selective estrogen receptor modulator (SERM) that is FDA-approved for treating dyspareunia related to VVA, and has shown superb improvements in overall sexual health. 104 women will be randomized to receive 12 weeks of 60mg oral ospemifene, taken daily, or 12 weeks of 0.5mg vaginal conjugated estrogens, which is placed vaginally twice per week. The improvements in sexual health and VVA symptom severity will be compared in each group. This study will help determine if ospemifene is a better treatment medication than conjugated estrogens.

DETAILED DESCRIPTION:
Female sexual dysfunction (FSD) affects 57% of postmenopausal women. Vulvovaginal atrophy (VVA) is a condition that impacts up to 60% of the growing postmenopausal female population, and the most common symptom is dyspareunia. Women with FSD are 3.84 times as likely to also have VVA. Vaginal estrogen is the most common treatment for VVA, but it only marginally improves overall sexual function, and many women and clinicians avoid using it because of the risks of exogenous estrogen use during menopause. Ospemifene is a non-estrogen selective estrogen receptor modulator (SERM) that is FDA-approved for treating dyspareunia related to VVA, and has shown superb improvements in overall sexual health. This oral medication, taken daily, improves vaginal health, and has demonstrated protective activity in the breast and bone tissues. It also has not demonstrated any carcinogenic activity in the endometrium or liver. This study hopes to determine if ospemifene is superior to conjugated estrogens in improving sexual function and vaginal atrophy symptoms.

104 women will be randomized to receive 12 weeks of 60mg oral ospemifene, taken daily, or 12 weeks of 0.5mg vaginal conjugated estrogens, which is placed vaginally twice per week. Each participant will be informed of her assigned medication, and will receive a medication coupon to help offset the cost of the medication. Each medication is FDA-approved for long-term use of at least 52 weeks. For this study, a 12-week prescription for the medication will be sent electronically to the pharmacy of the participant's choice. The improvements in sexual health and VVA symptom severity will be compared in each group.

ELIGIBILITY:
Inclusion Criteria:

* Interested in resuming or continuing sexual activity
* Greater than 12 months since last menstrual cycle or prior bilateral oophorectomy
* Dyspareunia as a vulvovaginal atrophy symptom
* Normal mammogram within 12 months prior to entry into the study

Exclusion Criteria:

* History or suspicion of breast carcinoma
* History of hormone-dependent tumor
* Genital bleeding of unknown cause
* Ongoing vaginal infection
* History of cerebrovascular accident (CVA), myocardial infarction (MI) or heart disease
* Uncontrolled hypertension (HTN) over 160/100
* Serious disease or chronic condition that may prevent completion of study
* Body Mass Index (BMI) over 40
* Hypercoagulable state, or currently on anticoagulant therapy
* Use of any exogenous sex hormone within three months from study entry, or during the study
* Pelvic surgery within the last 12 months

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Northington, MD, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Midtown Hospital, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory Hospital, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between June 2017 and September 2017
Pre-assignment Details: One individual gave informed consent to participate in the study and was randomized to the Estrogen arm.
Groups:
- Ospemifene: Women randomized to this arm were to receive 60mg oral ospemifene, taken daily, for 12 weeks
- Estrogen: Women randomized to this arm were to receive 0.5mg vaginal conjugated estrogens, placed vaginally twice per week, for 12 weeks
Period: Overall Study
Arm/Group | Ospemifene | Estrogen
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants consenting to take part in the trial are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ospemifene | Estrogen | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 51 (0.0) | 51 (0.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 1 | 1
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Female Sexual Function Index Score
Description: The Female Sexual Function Index (FSFI) is a 19 item questionnaire that asks about sexual function in the prior four weeks. The FSFI was developed for the specific purpose of assessing sexual arousal, orgasm, satisfaction, pain related to sexual functioning in clinical trial participants. Participants answer by selecting between 5-6 question-specific options to rate the degree to which the question fits their experience. Each response option is assigned a point and each question has 0-5 or 1-5 possible points. The points are summed to determine a total score. The total score can range from 2 to 36 and scores equal to or less than 26.55 indicate female sexual dysfunction (FSD).
Time Frame: Baseline, Week 12
Population: The single participant was lost to follow up prior to completing the Week 12 assessment.
Measure: Number; unit: units on a scale
Groups:
- Estrogen: Women randomized to this arm received 0.5mg vaginal conjugated estrogens, placed vaginally twice per week, for 12 weeks
Arm/Group | Estrogen
Number analyzed (Participants) | 1
units on a scale
  Baseline | 9
  Week 12: number analyzed (Participants) | 0

2. Primary Outcome: Pain With Sex
Description: Participants reported pain with sex at the Baseline Visit and after 12 weeks of treatment. Participants rated the severity of their symptoms from 0 to 3, where 0 = none, 1 = mild, 2 = moderate and 3 = severe.
Time Frame: Baseline, Week 12
Population: The single participant was lost to follow up prior to completing the Week 12 assessment.
Measure: Number; unit: units on a scale
Arm/Group | Estrogen
Number analyzed (Participants) | 1
units on a scale
  Baseline | 2
  Week 12: number analyzed (Participants) | 0

3. Primary Outcome: Vaginal Dryness
Description: Participants reported vaginal dryness at the Baseline Visit and after 12 weeks of treatment. Participants rated the severity of their symptoms from 0 to 3, where 0 = none, 1 = mild, 2 = moderate and 3 = severe.
Time Frame: Baseline, Week 12
Population: The single participant was lost to follow up prior to completing the Week 12 assessment.
Measure: Number; unit: units on a scale
Arm/Group | Estrogen
Number analyzed (Participants) | 1
units on a scale
  Baseline | 3
  Week 12: number analyzed (Participants) | 0

4. Primary Outcome: Vaginal Itching
Description: Participants reported vaginal itching at the Baseline Visit and after 12 weeks of treatment. Participants rated the severity of their symptoms from 0 to 3, where 0 = none, 1 = mild, 2 = moderate and 3 = severe.
Time Frame: Baseline, Week 12
Population: The single participant was lost to follow up prior to completing the Week 12 assessment.
Measure: Number; unit: units on a scale
Arm/Group | Estrogen
Number analyzed (Participants) | 1
units on a scale
  Baseline | 3
  Week 12: number analyzed (Participants) | 0

5. Primary Outcome: Vaginal Irritation
Description: Participants reported vaginal irritation at the Baseline Visit and after 12 weeks of treatment. Participants rated the severity of their symptoms from 0 to 3, where 0 = none, 1 = mild, 2 = moderate and 3 = severe.
Time Frame: Baseline, Week 12
Population: The single participant was lost to follow up prior to completing the Week 12 assessment.
Measure: Number; unit: units on a scale
Arm/Group | Estrogen
Number analyzed (Participants) | 1
units on a scale
  Baseline | 3
  Week 12: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the participant consented to take part in the study through the Week 12 Visit.
Arm/Group | Estrogen
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The patient population did not provide as many interested and qualified subjects as anticipated, thus the study was terminated early due to obstacles with recruitment and time limitations for data analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT03018106/Prot_SAP_000.pdf